CLINICAL TRIAL: NCT03900728
Title: Auriculotherapy as an Adjunct for Pain Management During Medication Abortion: a Randomized, Double-blinded, Three-arm Trial
Brief Title: Auriculotherapy During Medication Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Carolyn Westhoff, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AAAS2520
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Abortion Early
MeSH Terms: interventions — Auriculotherapy; Needles

STUDY DESIGN:
Intervention Model Description: This 3-arm randomized trial will assign participants 1:1:1 to receive either of two active treatments (acupuncture or acupressure) or placebo (insert adhesive disks applied to ears).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A separate investigator will apply the intervention after the initial usual care is complete and participants will go home using the intervention; thus the care provider will not be aware of the treatment. The adhesive disks appear similar for the treatments and the placebo arm; thus the participants will be unaware of their treatment assignment. The research assistant collecting the outcomes data will not know which treatment arm the participant belongs to. Finally, treatment assignment will be coded in the study database until analysis is complete, so that the investigator will be unaware of the treatment assignment until analysis is complete and then un-blinding will occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Auriculotherapy with needles (acupuncture) + usual care (Active Comparator): A designated trained therapist will perform auriculotherapy with 1mm (Pyonex) needles at five acupoints on each ear (10 points total). The needles are affixed with a small round adhesive disk. The needles will stay in place until removal at the 1-week follow-up visit
  Interventions: Device: Auriculotherapy with needles
- Auriculotherapy with gold beads (acupressure) + usual care (Active Comparator): A designated trained therapist will perform auriculotherapy with beads at five acupoints on each ear (10 points total). The beads are affixed with a small round adhesive disk. The beads will stay in place until removal at the 1-week follow-up visit.
  Interventions: Device: Auriculotherapy with beads
- Placebo group + usual care (Sham Comparator): A designated trained therapist will place adhesive disks at five acupoints on each ear (10 points total). The disks resemble those used with the active treatments. The disks will stay in place until removal at the 1-week follow-up visit.
  Interventions: Device: Placebo Adhesive disks

INTERVENTIONS:
Device: Auriculotherapy with needles — Single-use 1.2mm acupuncture press needles attach to pre-specified acupoints on the participant's ears with adhesive disk/tape.
  Other Names: Pyonex needles
  Arms: Auriculotherapy with needles (acupuncture) + usual care
Device: Auriculotherapy with beads — A trained co-investigator will place the beads onto prespecified acupoints of the participant's ears. An adhesive disk will adhere the beads to the ears.
  Other Names: Single-use gold-plated 1.2mm beads/balls attach to pre-specified acupoints on the participant's ears with adhesive disk/tape.
  Arms: Auriculotherapy with gold beads (acupressure) + usual care
Device: Placebo Adhesive disks — Single-use adhesive disks without needles or beads.
  Other Names: Placebo disks
  Arms: Placebo group + usual care

SUMMARY:
This randomized trial will evaluate the effect of adding auriculotherapy (i.e. acupuncture applied to the ear) using either gold beads or Pyonex needles in addition to usual care for the relief of pain and anxiety during medication abortion. The control group will receive placebo auriculotherapy plus usual care. Participants will receive the assigned treatment immediately after they receive their initial abortion medication. The investigators will assess pain and anxiety via text message once daily for four days, and in person at a one-week follow-up visit.

DETAILED DESCRIPTION:
Most women undergoing medication abortion with mifepristone and misoprostol report moderate to severe pain, despite treatment with ibuprofen or opioids. In 2018 National Academies of Sciences, Engineering and Medicine (NASEM) recommended research to improve pain relief. Limited data indicate that acupuncture is valuable for dysmenorrhea and for labor pain, conditions in which pain may be similar to that experienced during medication abortion. This randomized trial will recruit women seeking medication abortion after they have completed their routine clinical assessment and after they have received mifepristone. This study will evaluate two types of auriculotherapy applied to selected acupoints on the external ear. The study treatments are acupuncture using Pyonex needles and acupressure using gold pellets; both are applied to the ear using adhesive disks. A control group will receive the adhesive disks alone. All participants will receive usual medication abortion care, including taking misoprostol 1-3 days after mifepristone and ibuprofen for pain management. The investigators will query the participants regarding pain and anxiety. Follow-up will end at the time of the usual clinical follow-up about one week after mifepristone administration.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant up to 10 weeks (70 days) gestation
* Seeking medication abortion with mifepristone and misoprostol
* Initial clinical care completed and mifepristone administered
* English- or Spanish-speaking
* Able to use a mobile phone for follow-up on days 1-4

Exclusion Criteria:

* Not a candidate for medication abortion for any reason
* Allergy to adhesives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 138 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, Principal Investigator — Coumbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Absent personal identifiers, we will share pain and anxiety outcome data with researchers carrying out similar trials in order to conduct individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after acceptance of main study outcome paper for publication.
Access Criteria: By personal contact with PI

REFERENCES:
- [Background] Ndubisi C, Danvers A, Gold MA, Morrow L, Westhoff CL. Auricular acupuncture as an adjunct for pain management during first trimester abortion: a randomized, double-blinded, three arm trial. Contraception. 2019 Mar;99(3):143-147. doi: 10.1016/j.contraception.2018.11.016. Epub 2018 Dec 7. PMID 30529393
- [Result] Westhoff CL, Nelson IS, Suarez-Rodriguez A, Gold MA. Auricular acupressure and acupuncture as adjuncts for pain management during first trimester medication abortion: A randomized three-arm trial. Contraception. 2021 May;103(5):348-355. doi: 10.1016/j.contraception.2020.12.003. Epub 2020 Dec 17. PMID 33340496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 138 enrolled subjects, 2 subjects were not randomized. 1 subject did not have a study auriculotherapist available during the visit and 1 subject declined randomization. Only data information for the randomized subjects were analyzed (n = 136).
Period: Overall Study
Arm/Group | Auriculotherapy With Needles (Acupuncture) + Usual Care | Auriculotherapy With Gold Beads (Acupressure) + Usual Care | Placebo Group + Usual Care
Started | 40 | 57 | 39
Completed | 40 | 57 | 35
Not Completed | 0 | 0 | 4
Not completed — No text responses | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auriculotherapy With Needles (Acupuncture) + Usual Care | Auriculotherapy With Gold Beads (Acupressure) + Usual Care | Placebo Group + Usual Care | Total
Number analyzed (Participants) | 40 | 57 | 39 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (5.8) | 28.6 (7.0) | 27.3 (5.9) | 27.67 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 57 | 39 | 136
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 51 | 35 | 121
  Not Hispanic or Latino | 5 | 6 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 57 | 39 | 136

OUTCOME MEASURES:

1. Primary Outcome: Pain VAS Score
Description: Self-assessed maximum pain reported using a 0-100 mm visual analog scale (VAS), where 100 signifies maximum pain.
Time Frame: Auriculotherapy is applied on the day of mifepristone. Participants take misoprostol 1-3 days later. Pain scores are recorded following misoprostol at 8pm x 4 days (selecting the highest of the 4 for analysis).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Auriculotherapy With Needles (Acupuncture) + Usual Care | Auriculotherapy With Gold Beads (Acupressure) + Usual Care | Placebo Group + Usual Care
Number analyzed (Participants) | 40 | 57 | 39
score on a scale | 75 [45 to 90] | 60 [20 to 85] | 55 [30 to 85]

2. Secondary Outcome: Anxiety VAS Score
Description: Self-assessed maximum anxiety reported using a 0-100 mm visual analog scale, where 100 signifies maximum anxiety.
Time Frame: Auriculotherapy is applied on the day of mifepristone. Participants take misoprostol 1-3 days later. Anxiety scores are recorded following misoprostol at 8pm x 4 days (selecting the highest of 4 for analysis).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Auriculotherapy With Needles (Acupuncture) + Usual Care | Auriculotherapy With Gold Beads (Acupressure) + Usual Care | Placebo Group + Usual Care
Number analyzed (Participants) | 40 | 57 | 39
score on a scale | 45 [0 to 60] | 10 [0 to 50] | 30 [0 to 50]

ADVERSE EVENTS:
Time Frame: Up to 1 week post administration
Arm/Group | Auriculotherapy With Needles (Acupuncture) + Usual Care | Auriculotherapy With Gold Beads (Acupressure) + Usual Care | Placebo Group + Usual Care
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/57 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/57 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/57 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT03900728/Prot_SAP_000.pdf